CLINICAL TRIAL: NCT03614962
Title: Efficacy of Warmth and Transcutaneous Electrical Nerve Stimulation (TENS) in Improving Cognitive Functions and Behavioral Symptoms in Older Adults with Dementia: a Randomized, Controlled Clinical Trial
Brief Title: Warmth and Transcutaneous Electrical Nerve Stimulation (TENS) in Improving Cognitive Functions in People with Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Shamay Ng, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018_ITF_MRP
Record Dates: First submitted 2018-07-15; First posted 2018-08-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Dementia
Keywords: Transcutaneous electrical nerve stimulation; Cognitive; Memory
MeSH Terms: conditions — Dementia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Warmth + TENS group (Experimental): All participants will be offered a hat device that elicits warmth and TENS.
  Interventions: Device: Warmth + TENS
- Warmth + placebo-TENS group (Active Comparator): All participants will be offered a hat device that elicits warmth and placebo-TENS.
  Interventions: Device: Warmth + placebo-TENS
- Warmth group (Active Comparator): All participants will be offered a hat device that elicits warmth only.
  Interventions: Device: Warmth only
- TENS group (Active Comparator): All participants will be offered a hat device that elicits TENS only.
  Interventions: Device: Warmth + TENS; Device: TENS
- control group (Sham Comparator): All participants will be offered a hat device that without warmth or TENS output.
  Interventions: Device: control

INTERVENTIONS:
Device: Warmth + TENS — A hat device will offer the electrical stimulation (pulse width of 120 milliseconds at about 100 Hz with constant current 0.02mA-0.7 mA, intensity setting at sensory threshold) over 4 acupuncture points over the scalp, including Baihui (GV20), Sishencong (EX-HN1), Fengchi (GB20) and Shenting (GV24). Selection of acupuncture points has been based on the recommendation of traditional Chinese medicine.
  A custom-built warmth pad surrounding the TENS electrodes could produce the controlled comfortable warmth sensation, with default setting at 37degrees to 40 degrees Celsius.
  Arms: TENS group; Warmth + TENS group
Device: Warmth + placebo-TENS — A custom-built warmth pad surrounding the TENS electrodes could produce the controlled comfortable warmth sensation, with default setting at 37degrees to 40 degrees Celsius. The TENS electrodes are presented in the cap but no output will be delivered via these electrodes.
  Arms: Warmth + placebo-TENS group
Device: TENS — A hat device will offer the electrical stimulation (pulse width of 120 milliseconds at about 100 Hz with constant current 0.02mA-0.7 mA, intensity setting at sensory threshold) over 4 acupuncture points over the scalp, including Baihui (GV20), Sishencong (EX-HN1), Fengchi (GB20) and Shenting (GV24). Selection of acupuncture points has been based on the recommendation of traditional Chinese medicine.
  Arms: TENS group
Device: Warmth only — A custom-built warmth pad surrounding the TENS electrodes could produce the controlled comfortable warmth sensation, with default setting at 37degrees to 40 degrees Celsius. No built-in TENS electrodes in the cap.
  Arms: Warmth group
Device: control — No warmth pad and TENS electrodes presented in the cap.
  Arms: control group

SUMMARY:
Evidence showed that both TENS and passive body heating are potential treatment strategies for improving cognitive functions in people with dementia. It is hypothesized that hat device (Warmth +TENS) over the 4 acupuncture points would induce a greater improvement in cognitive functions and behavioural symptoms when compared with other hat devices (Warmth + placebo-TENS; TENS only; Warmth alone) and Control (hat device with no warmth and no TENS).

DETAILED DESCRIPTION:
Acupuncture, a primary therapeutic method in traditional Chinese medicine, has been used for patients with dementia to improve memory, orientation, calculation, and self-managing ability in patients having dementia and prevent decline of cognitive functions. Results of animal studies have demonstrated that electroacupuncture on the head region is effective in managing the symptoms associated with dementia, including vascular dementia.

A review of 8 studies on effects of TENS on non-pain related cognitive and behavioural functioning in patients with Alzheimer's disease and non-demented patients concluded that TENS could improve memory, affective behaviour and rest-activity rhythm in patients having Alzheimer's disease.

Passive body heating is another novel physical intervention strategy which potentially can relieve the symptoms of dementia. A previous study demonstrated that the attention function of 15 elderly, measured by the reaction time in the Rapid Visual Processing Test, improved after passive body heating via a thermal suit. Moreover, 30 minutes of hot-water immersion improved the sleep quality in 13 people with vascular dementia.

ELIGIBILITY:
Inclusion Criteria:

1. are currently diagnosed having Alzheimer's disease, vascular dementia or mixed-type mild to major neurocognitive disorder based on the Fifth Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM -5) by psychogeriatrician with more than 3 years of experience in dementia diagnosis;
2. are categorized in the mild or moderate degree of dementia based on the Global Deterioration Scale;
3. have a stable drug intake for the past 3 months;
4. live with at least 1 caregiver in the community;
5. are able to follow simple instructions;
6. are able to give informed consent by them or their family members.

Exclusion Criteria:

1. have unstable medical conditions or severe behavioural disturbances, which do not allow participation in the study as judged by the study psychogeriatrician,
2. have any additional medical, cardiovascular , orthopedic or cognitive conditions, such as having uncontrolled hypertension unstable angina and comorbid schizophrenia, that would hinder proper assessment and treatment.
3. use a cardiac pacemaker,
4. live in old age home, elderly home or care and attention homes,
5. receive long term nursing home placements of patients during the treatment phase

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
The Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) - Baseline | Baseline (0 week)
  The HK-MoCA will be used to assess the level of cognitive impairment. The scores of HK-MoCA ranging from 0 to 30, with a higher score indicates a higher level of cognitive function. This instrument was designed to evaluate 7 domains of cognitive functions which are key determinants of the functional performance of the participants, namely visuospatial/executive functions, naming, verbal memory registration and learning, attention, abstraction, delayed verbal memory.
The Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) - post intervention | 6 weeks
  The HK-MoCA will be used to assess the level of cognitive impairment. The scores of HK-MoCA ranging from 0 to 30, with a higher score indicates a higher level of cognitive function. This instrument was designed to evaluate 7 domains of cognitive functions which are key determinants of the functional performance of the participants, namely visuospatial/executive functions, naming, verbal memory registration and learning, attention, abstraction, delayed verbal memory.
The Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) - short term followup | 10 weeks
  The HK-MoCA will be used to assess the level of cognitive impairment. The scores of HK-MoCA ranging from 0 to 30, with a higher score indicates a higher level of cognitive function. This instrument was designed to evaluate 7 domains of cognitive functions which are key determinants of the functional performance of the participants, namely visuospatial/executive functions, naming, verbal memory registration and learning, attention, abstraction, delayed verbal memory.
The Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) - long term followup | 62 weeks
  The HK-MoCA will be used to assess the level of cognitive impairment. The scores of HK-MoCA ranging from 0 to 30, with a higher score indicates a higher level of cognitive function. This instrument was designed to evaluate 7 domains of cognitive functions which are key determinants of the functional performance of the participants, namely visuospatial/executive functions, naming, verbal memory registration and learning, attention, abstraction, delayed verbal memory.

SECONDARY OUTCOMES:
Chinese version of Disability Assessment for Dementia (C-DAD) - baseline | baseline (0 week)
  C-DAD will be used to assess the participant's ability to perform a spectrum of functional activities, such as going on an outing and housekeeping. During the assessment, a caregiver is asked to indicate if the participant was able to perform 47 daily activities within the previous weeks with the responses of 'yes', ''no' or 'not applicable'. The result will then be converted into a scale ranging from 0 to 100, with a higher score indicates a higher level of functioning.
Chinese version of Disability Assessment for Dementia (C-DAD) - post intervention | 6 weeks
  C-DAD will be used to assess the participant's ability to perform a spectrum of functional activities, such as going on an outing and housekeeping. During the assessment, a caregiver is asked to indicate if the participant was able to perform 47 daily activities within the previous weeks with the responses of 'yes', ''no' or 'not applicable'. The result will then be converted into a scale ranging from 0 to 100, with a higher score indicates a higher level of functioning.
Chinese version of Disability Assessment for Dementia (C-DAD) - short term followup | 10 weeks
  C-DAD will be used to assess the participant's ability to perform a spectrum of functional activities, such as going on an outing and housekeeping. During the assessment, a caregiver is asked to indicate if the participant was able to perform 47 daily activities within the previous weeks with the responses of 'yes', ''no' or 'not applicable'. The result will then be converted into a scale ranging from 0 to 100, with a higher score indicates a higher level of functioning.
Chinese version of Disability Assessment for Dementia (C-DAD) - long term followup | 62 weeks
  C-DAD will be used to assess the participant's ability to perform a spectrum of functional activities, such as going on an outing and housekeeping. During the assessment, a caregiver is asked to indicate if the participant was able to perform 47 daily activities within the previous weeks with the responses of 'yes', ''no' or 'not applicable'. The result will then be converted into a scale ranging from 0 to 100, with a higher score indicates a higher level of functioning.
Pittsburg Sleep Quality Index (PSQI) - baseline | baseline (0 weeks)
  PSQI will be used to assess the participant's sleep quality for the past months. PSQI consists of 19 individual items including sleep duration, sleep latency, sleep disturbance etc. The total score will be range from 0-21 and lower scores indicate a better sleep quality.
Pittsburg Sleep Quality Index (PSQI) - post intervention | 6 weeks
  PSQI will be used to assess the participant's sleep quality for the past months. PSQI consists of 19 individual items including sleep duration, sleep latency, sleep disturbance etc. The total score will be range from 0-21 and lower scores indicate a better sleep quality.
Pittsburg Sleep Quality Index (PSQI) - short term followup | 10 weeks
  PSQI will be used to assess the participant's sleep quality for the past months. PSQI consists of 19 individual items including sleep duration, sleep latency, sleep disturbance etc. The total score will be range from 0-21 and lower scores indicate a better sleep quality.
Pittsburg Sleep Quality Index (PSQI) - long term followup | 62 weeks
  PSQI will be used to assess the participant's sleep quality for the past months. PSQI consists of 19 individual items including sleep duration, sleep latency, sleep disturbance etc. The total score will be range from 0-21 and lower scores indicate a better sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: SSM Ng, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong